CLINICAL TRIAL: NCT00134043
Title: Phase II Study of Histone Deacetylase Inhibitor SAHA (Vorinostat) in Patients With Metastatic Thyroid Carcinoma
Brief Title: Suberoylanilide Hydroxamic Acid in Treating Patients With Metastatic and/or Locally Advanced or Locally Recurrent Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01468; 04110; CDR0000439450; NCI-6902; OSU-04110; N01CM62207 (NIH)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Insular Thyroid Cancer; Recurrent Thyroid Cancer; Stage II Follicular Thyroid Cancer; Stage II Papillary Thyroid Cancer; Stage IV Follicular Thyroid Cancer; Stage IV Papillary Thyroid Cancer; Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Carcinoma, Medullary | interventions — Vorinostat

ARMS (1):
- Arm I (Experimental): Patients receive oral suberoylanilide hydroxamic acid (SAHA) twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are then evaluated for disease response. Patients achieving a complete response receive an additional 2 courses of SAHA. Patients achieving stable disease or a partial response receive 4 additional courses of SAHA.After completion of study treatment, patients are followed within 4 weeks.
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza

SUMMARY:
This phase II trial is studying how well suberoylanilide hydroxamic acid works in treating patients with metastatic and/or locally advanced or locally recurrent thyroid cancer. Drugs used in chemotherapy, such as suberoylanilide hydroxamic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Suberoylanilide hydroxamic acid may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with metastatic and/or locally advanced or locally recurrent thyroid cancer treated with suberoylanilide hydroxamic acid.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this drug in these patients.

OUTLINE:

Patients receive oral suberoylanilide hydroxamic acid (SAHA) twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are then evaluated for disease response. Patients achieving a complete response receive an additional 2 courses of SAHA. Patients achieving stable disease or a partial response receive 4 additional courses of SAHA. After completion of study treatment, patients are followed within 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed thyroid cancer

  * One of the following subtypes:

    * Papillary thyroid cancer
    * Follicular thyroid cancer
    * Hürthle cell thyroid cancer
    * Insular thyroid cancer
    * Medullary thyroid cancer
    * Mixed histology thyroid cancer
    * Poorly differentiated thyroid cancer
    * Tall-cell thyroid cancer
  * Metastatic and/or locally advanced or locally recurrent disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Lesions in a previously irradiated area allowed provided there has been subsequent disease progression of the irradiated lesions
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* Not a candidate for radioactive iodine I^131 therapy
* Performance status - ECOG 0-1
* At least 6 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drug
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No other active malignancy except nonmetastatic nonmelanoma skin cancer or carcinoma in situ of the cervix
* More than 4 weeks since prior systemic cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No more than 2 prior chemotherapy regimens for the treatment of thyroid cancer
* See Disease Characteristics
* More than 4 weeks since prior external beam radiotherapy
* At least 24 weeks since prior radioactive iodine I^131 therapy
* Recovered from prior therapy
* More than 4 weeks since prior valproic acid or any other histone deacetylase inhibitor
* More than 4 weeks since prior investigational tumor-specific therapy
* Concurrent oral or IV bisphosphonates for bony metastases allowed at the discretion of the investigator
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent tumor-specific or investigational therapy
* No other concurrent anticancer therapy
* No concurrent adjuvant therapy for another cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Woyach JA, Kloos RT, Ringel MD, Arbogast D, Collamore M, Zwiebel JA, Grever M, Villalona-Calero M, Shah MH. Lack of therapeutic effect of the histone deacetylase inhibitor vorinostat in patients with metastatic radioiodine-refractory thyroid carcinoma. J Clin Endocrinol Metab. 2009 Jan;94(1):164-70. doi: 10.1210/jc.2008-1631. Epub 2008 Oct 14. PMID 18854394

RESULTS

PARTICIPANT FLOW:
Groups:
- DTCs (Well-differentiated Thyroid Carcinomas); MTC (Medullary Thyroid Cancer): Patients receive oral suberoylanilide hydroxamic acid (SAHA) twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are then evaluated for disease response. Patients achieving a complete response receive an additional 2 courses of SAHA. Patients achieving stable disease or a partial response receive 4 additional courses of SAHA.After completion of study treatment, patients are followed within 4 weeks.
  vorinostat: Given orally
Period: Overall Study
Arm/Group | DTCs (Well-differentiated Thyroid Carcinomas) | MTC (Medullary Thyroid Cancer)
Started | 16 | 3
Completed | 16 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTCs (Well-differentiated Thyroid Carcinomas) | MTC (Medullary Thyroid Cancer) | Total
Number analyzed (Participants) | 16 | 3 | 19
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 77] | 65 [54 to 67] | 64 [40 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 12
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 13 | 3 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 3 | 18
  Canada | 1 | 0 | 1
ECOG (Eastern Cooperative Oncology Group) performance status [Number; unit: participants]
  0 (Fully active) | 6 | 2 | 8
  1(restricted in physically strenuous activity) | 10 | 1 | 11
Site of metastasis [Number; unit: participants]
  Lungs | 16 | 0 | 16
  Lymph nodes | 8 | 1 | 9
  Bones | 4 | 2 | 6
  Brain | 4 | 0 | 4
  1-2 sites | 13 | 1 | 14
  More than 2 sites | 3 | 2 | 5
Previous therapies [Number; unit: number of]
  Surgery | 15 | 3 | 18
  Iodin-131 | 16 | 0 | 16
  External beam radiation | 6 | 2 | 8
  Cytotoxic chemotherapy | 6 | 2 | 8
Pathology of thyroid carcinoma [Number; unit: participants]
  Classic PTC | 12 | 0 | 12
  Follicular variant of PTC | 2 | 0 | 2
  FTC | 1 | 0 | 1
  Hurthle cell | 1 | 0 | 1
  MTC | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (PR + CR) Using RECIST/WHO Response Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: Up to 3 years
Population: Per RECIST (Response Evaluation Criteria in Solid Tumors)
Measure: Number; unit: percentage of participants
Groups:
- DTCs (Well-differentiated Thyroid Carcinomas): Patients receive oral suberoylanilide hydroxamic acid (SAHA) twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are then evaluated for disease response. Patients achieving a complete response receive an additional 2 courses of SAHA. Patients achieving stable disease or a partial response receive 4 additional courses of SAHA.After completion of study treatment, patients are followed within 4 weeks.
Arm/Group | DTCs (Well-differentiated Thyroid Carcinomas) | MTC (Medullary Thyroid Cancer)
Number analyzed (Participants) | 16 | 5
percentage of participants
  PR (Partial Response) | 0 | 0
  CR (Complete Response) | 0 | 0
  Stable disease | 56 | 0

ADVERSE EVENTS:
Time Frame: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was utilized for adverse event reporting.
Description: AEs were worst grade experienced by patient on study and were primarily grade 1-3 according to the NCI Common Terminology Criteria for Adverse Events version 3.0
Groups:
- Arm I & Arm II: Patients receive oral suberoylanilide hydroxamic acid (SAHA) twice daily on days 1-14. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are then evaluated for disease response. Patients achieving a complete response receive an additional 2 courses of SAHA. Patients achieving stable disease or a partial response receive 4 additional courses of SAHA.After completion of study treatment, patients are followed within 4 weeks.
  vorinostat: Given orally
Arm/Group | Arm I & Arm II
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 19/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I & Arm II (N=19)
Abdominal Cramping (Gastrointestinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 16 (16)
Anxiety (Psychiatric disorders) | 1 (1)
Arterial thrombus (Vascular disorders) | 1 (1)
Ataxia (Nervous system disorders) | 3 (3)
Blurry vision (Eye disorders) | 2 (2)
Bronchitis/pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bruising/hematoma (Vascular disorders) | 3 (3)
Chest pain (muscle) (General disorders) | 3 (3)
Chills/Sweating (General disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Dizziness (Nervous system disorders) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 5 (5)
Dsypnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 15 (15)
Flatulence/Bloating (Gastrointestinal disorders) | 6 (6)
Flushing (Vascular disorders) | 2 (2)
General Weakness (Musculoskeletal and connective tissue disorders) | 7 (7)
General pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Heartburn (Gastrointestinal disorders) | 3 (3)
Herpes zoster (Investigations) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Memory loss (Nervous system disorders) | 3 (3)
Minor bleeding (Vascular disorders) | 5 (5)
Mouth sores (Gastrointestinal disorders) | 4 (4)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 5 (5)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea/Vomiting (Gastrointestinal disorders) | 13 (13)
Paresthesias (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Taste changes (Gastrointestinal disorders) | 9 (9)
Tremor (Nervous system disorders) | 2 (2)
Weight loss (Investigations) | 13 (13)
Anemia (Blood and lymphatic system disorders) | 15 (15)
Leukopenia (Blood and lymphatic system disorders) | 12 (12)
Neutropenia (Investigations) | 7 (7)
Lymphopenia (Investigations) | 2 (2)
Thrombocytopenia (Injury, poisoning and procedural complications) | 14 (14)
High PTT (Investigations) | 2 (2)
High P/INR (Investigations) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less